CLINICAL TRIAL: NCT03986229
Title: Evaluation of the Effect of Custom Compression Garments on Standing Static Balance in Ehlers Danlos Syndrome
Acronym: EDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/18/0360
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Ehlers-Danlos Syndrome
Keywords: ehlers-danlos syndrome; static balance; custom compression garments
MeSH Terms: conditions — Ehlers-Danlos Syndrome

STUDY DESIGN:
Intervention Model Description: 15 patients exposed to the AB sequence and 15 patients exposed to the BA sequence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With compression garments (Active Comparator): Evaluation of the variation in the travel speed of the "center of pressure" with compression garments and the standing static balance.
  Interventions: Other: Evaluate the variation in the travel speed of the "center of pressure" with and without compression garments.
- Without compression garments (Active Comparator): Evaluation of the variation in the travel speed of the "center of pressure" with compression garments and the standing static balance.
  Interventions: Other: Evaluate the variation in the travel speed of the "center of pressure" with and without compression garments.

INTERVENTIONS:
Other: Evaluate the variation in the travel speed of the "center of pressure" with and without compression garments. — Each evaluation will be done according to the following protocol:
  * Evaluation of the pain
  * Berg test
  * One test per condition starting with open eyes
  * Standardized instructions:
  * Break about 15 minutes (wash-out) between each test.
  * Both conditions will be tested on the same day.
  * Evaluation in an environment free from visual and audible interference.

SUMMARY:
Studies have shown the existence of a proprioceptive deficit in patients with Ehlers Danlos Syndrome (EDS) (genetic pathology of connective tissue with hypermobility, multifactor joint instability). A study dating from 2010 showed a qualitative improvement in disability when wearing compression garments (CG) in this pathology, particularly in the fields of proprioception and balance.

The purpose of this study is to quantify the effect of CG on standing static balance in patients with EDS.

DETAILED DESCRIPTION:
To evaluate the effect of CG on standing static balance in patients with EDS, this study is a pilot study, carried out according to a cross-over scheme of type AB/BA.

Each patient will benefit from 2 posturological evaluations, namely without CG (treatment A) and with CG (treatment B). Patients will be randomly assigned to 2 groups: the AB or BA sequence will be randomized for each patient.

For each evaluation, a measurement with eyes open and eyes closed will be performed.

A clinical balance assessment by the Berg test will be performed for each of the conditions.

ELIGIBILITY:
Inclusion Criteria:

* EDS patients over 18 years of age walking around without technical assistance.
* Patients will need to be diagnosed both during the interview (presence of a family history, hypermobility and joint instability that has been evolving for years) and with a guide for analysis from EDS to AP-HP.
* Beighton's score must be 5/9 or higher.
* Free from any other pathology likely to have an impact on the balance.
* Patient with a CG as part of his or her management of the EDS
* Sufficient understanding to understand the objectives of the study and give consent.
* Patient affiliated or benefiting from a social security scheme
* Allergies to one of the components (Polyamide and Elastane) of the CG
* Recent compression garments less than 6 months old.

Exclusion Criteria:

* Patient under guardianship, curators, justice protection.
* Comorbidity likely to influence balance.
* Significant pain (assessed by the patient) induced by the use of CG.
* Any acute event requires the postponement of the assessment to ensure that the patient's progress is in the usual conditions.
* Any acute pathology having an impact on the musculoskeletal system and/or general condition.
* Pregnancy/breastfeeding
* Compression garments over 6 months old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Evaluate the variation in the travel speed of the "center of pressure" (COP) with compression garments | 15 minutes
  Each patient will benefit from 2 posturological evaluations, namely without CG (treatment A) and with CG (treatment B).
Evaluate the variation in the travel speed of the "center of pressure" without compression garments. | 30 minutes
  Evaluate the variation in the travel speed of the "center of pressure" without compression garments. Each patient will benefit from 2 posturological evaluations, namely without CG (treatment A) and with CG (treatment B).

SECONDARY OUTCOMES:
Evaluate the amplitude of the antero-posterior and lateral oscillations without compression garments | 15 minutes
  Evaluate the amplitude of the antero-posterior and lateral oscillations of the COP with and without compression garments Compare the stabilometric data with a clinical trial evaluating the reference balance.
Evaluate the amplitude of the antero-posterior and lateral oscillations without compression garments | 30 minutes
  Evaluate the amplitude of the antero-posterior and lateral oscillations of the COP with and without compression garments.
  Compare the stabilometric data with a clinical trial evaluating the reference balance.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Van Den Bossche, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Service de Medecine physique et réadaptation, Toulouse, Salies Du Salat, France

IPD SHARING:
Plan to Share IPD: No